CLINICAL TRIAL: NCT03742687
Title: HERAN-Heterogeneously Hypofractionated Radiotherapy for Locally Advanced NSCLC
Brief Title: Heterogeneously Hypofractionated Radiotherapy for Locally Advanced NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Lung Cancer Group (Other)
Collaborators: Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Vejle Hospital (Other); Herlev Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Azza A Khalil, Team leder, Consulant, MD, PhD, Danish Lung Cancer Group
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HERAN
Record Dates: First submitted 2017-10-11; First posted 2018-11-15 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Stage III Non-small-cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Radiotherapy Side Effect
Keywords: Locally advanced NSCLC; Radiotherapy; Hypofractionation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A:Large target volume (Experimental): The target volume for radiotherapy treatment volume is considered too large for a standard treatment of 66Gy in 33 fractions, considering the expected normal tissue toxicity with a standard treatment plan. Heterogeneously Hypofractionated Radiotherapy plan ( 24 fractions )
  Interventions: Radiation: Heterogeneously Hypofractionated Radiotherapy
- B:Fragile patient (Experimental): The patient is too fragile for standard long-course radiotherapy with 66 Gy. Heterogeneously Hypofractionated Radiotherapy plan ( 24 fractions )
  Interventions: Radiation: Heterogeneously Hypofractionated Radiotherapy

INTERVENTIONS:
Radiation: Heterogeneously Hypofractionated Radiotherapy — A heterogeneous hypofractionated schedule for the treatment of high-risk locally advanced NSCLC patients in which the central idea is to decrease dose to normal tissue by ascribing a heterogeneous dose to the PTV. The dose to the periphery of the PTV as well as to the majority of lymph node targets is decreased compared to a standard treatment. The gross volume of the primary tumour and bulky lymph nodes receive mean doses of up to 66 Gy in 24 fractions, and thus receive a hypofractionated higher biological effective dose than standard 66 Gy in 33 fractions.

SUMMARY:
The options for patients with locally advanced non-small cell lung cancer (NSCLC) who are not candidates for a standard definitive chemoradiotherapy regime are meagre. These are patients who are not fit for a chemoradiotherapy schedule of 66 Gy in 2 Gy fractions due to either tumour extent, resulting in excessive dose to the healthy tissue in the thorax, or with performance status not supporting seven weeks of intensive treatment.

The aim is to study the efficiency as well as the safety of a new treatment option of heterogeneously hypofractionated radiotherapy for patients with locally advanced NSCLC who are not candidates for standard, high-dose chemoradiotherapy, either due to excessive irradiation of normal tissue (defined as category A patients) or due to fragility of the patient (category B patients).

DETAILED DESCRIPTION:
1.1 Radiotherapy in lung cancer The options for patients with locally advanced non-small cell lung cancer (NSCLC) who are not candidates for a standard definitive chemoradiotherapy regime are meagre. These patients are not fit for a standard chemoradiotherapy due to either tumour extent, resulting in excessive dose to the healthy tissue in the thorax, or with performance status not supporting seven weeks of intensive treatment. Such patients could benefit from a treatment offering long-term locoregional control leading to improved survival. However, at present, they are offered palliative treatment regimens. Alternatively, a full schedule of definitive chemoradiotherapy is sometimes attempted, and patient may only complete part of the treatment course.

Favourable alternative treatment options for this group of patients would have to:

* Provide a reasonable probability of locoregional disease control.
* Result in less expected toxicity.
* Be delivered using a shorter treatment schedule than the current 6-7 weeks Standard chemoradiotherapy aims at delivering a homogeneous dose distribution to the primary tumour and involved lymph nodes. However, studies of patterns of failures in locally advanced NSCLC patients indicate that isolated mediastinal nodal failures are less common than disease recurrence in the primary tumour site or in bulky lymph nodes. This suggests that it might be possible to lower the dose to all or selected parts of the involved mediastinal lymph nodes without drastically impacting the combined locoregional control.

Modelling studies indicate that tumour control may mainly depend on mean tumour dose, provided that the minimum dose to the tumour exceeds a certain level. One example is provided by stereotactic radiotherapy (SBRT), where very heterogeneous dose distributions usually results in higher dose in the middle of the tumour compared to the dose to the tumour periphery. The Danish NARLAL2 trial [NCT02354274] investigates heterogeneous dose escalation; with the most PET-avid part of the tumour used as a driver for the dose escalation. Most prospective trials have focused on hyperfractionated, accelerated treatments. Although effective, these schedules are also associated with substantial acute toxicity, likely not tolerable for borderline curative patients with extensive local disease. Definitive moderately hypofractioned radiotherapy has limited clinical evidence in lung cancer patients, but has demonstrated promising outcomes in a few trials. The current study aims to use a heterogeneous hypofractionated schedule for the treatment of high-risk locally advanced NSCLC patients, in order to improve loco-regional control and survival. The central idea is to decrease dose to normal tissue by ascribing a heterogeneous dose to the PTV. The gross volume of the primary tumour and bulky lymph nodes receive mean doses of up to 66 Gy in 24 fractions, and thus receive a hypofractionated higher biological effective dose than standard 66 Gy in 33 fractions.

1.2 Aim of this study To study the efficiency as well as the safety of a new treatment option of heterogeneously hypofractionated radiotherapy for patients with locally advanced NSCLC who are not candidates for standard, high-dose chemoradiotherapy, either due to excessive irradiation of normal tissue (defined as category A patients) or due to fragility of the patient (category B patients).

2 Purpose To demonstrate the feasibility of a heterogeneous and hypo-fractionated definitive (chemo-) radiotherapy schedule for locally advanced non-small cell lung cancer patients not candidates for standard, long-course chemoradiotherapy. Outcomes will be reported using descriptive statistics, from which the viability of the regimen as a standard treatment will be evaluated.

3 Study design This is a prospective multicentre feasibility study. It includes patients with inoperable locally advanced NSCLC (stage IIB-IV) not candidates for standard treatment with curative intent. Patients are treated with (chemo-) radiotherapy in 24 fractions, 5 fractions a week.

3.1 Systemic therapy Patients are allowed to receive 1-2 cycles of induction therapy with platinum doublet and/or concomitant chemotherapy. Patients with synthesizing mutations such as EGFR or ALK are allowed to receive TKI either as induction or as concurrent according to the local institution's guidelines.

3.2 Study sample size and time frame Patients in Denmark with NSCLC treated with palliative intent in 2014 had a one-year overall survival of 37.5%. The study is expected to enrol patients over a 2-year period, calculated from the date where two centres have opened for enrolment. At least 76 patients from category A and at least 75 patients from category B 3.3 Continuous monitoring of early mortality Any patient death within the first three months of radiotherapy initiation will be evaluated by the local site investigator and reported to primary investigator. Primary investigator will provide continuous monitoring of early mortality in order to ensure that the rate is not unacceptable, and will provide reports to all investigators at regular intervals.

3.4 Data management All dose plans used for patient treatment, including adapted plans, are exported to the national dose plan bank (CIRRO), from where doses to tumour, lymph nodes and organs at risk are extracted for analysis.

Baseline PET-CT scans as well as any CT or PET-CT scans at time of disease recurrence should, if available, preferably also be transferred to the dose plan bank.

4 Radiotherapy treatment planning 4.1 Scan procedure

A CT scan taking into account respiratory motion (i.e. 4D-CT scan, deep inspiration breath hold CT scan, or other respiratory controlled CT scans) is acquired:

* With intravenous contrast if allowed by kidney function.
* Maximum 3 mm distance between CT slices.
* Less than four weeks before start of radiotherapy A FDG-PET scan acquired within six week of the planning-CT should be used to guide the target delineation.

4.2 Target volumes The primary tumour is delineated separately as GTV-T. GTV-N includes all pathological lymph nodes. In patients with bulky lymph nodes, the dose will be escalated to the bulky part of the lymph nodes only, delineated in a separate structure, GTV-Nhigh. Bulky lymph nodes are defined as lymph nodes or conglomerates of lymph nodes where the longest diameter is 3 cm or more, i.e. corresponding to minimum volume of 14 cm3 for an approximately spherical target.

4.3 Dose planning Patients are treated with intensity-modulated radiotherapy (static beam angles or arc technique). Modern dose calculation algorithms (Monte Carlo, AAA, Collapsed Cone or similar) must be used to account for inhomogeneity corrections. Margins are applied ensuring that CTV receives a minimum dose of 95% of 50 Gy. All treatments are delivered in 24 fractions, 5 fractions per week.

5 Treatment verification and quality assurance 5.1 Verification of treatment position Daily imaging must be performed and used for daily correction of treatment position. Tolerances and margins depend on the setup strategy and must be defined locally.

5.2 Adaptive strategy and tumour shrinkage For patients where either the position of the tumour, the position of the lymph nodes, patient anatomy, or lung density changes are observed to result in dosimetric or geometric changes above the clinic specific tolerances, the radiotherapy treatment plan has to be adapted to the observed changes. Deliberate reduction of treatment volumes due to tumour shrinkage, is not encouraged.

5.3 Quality assurance To achieve similar dose planning strategies, all initially participating centres have performed dose planning for two representative patients. Centres joining the protocol will plan the same patients before including patients for comparison. Those plans are to be evaluated by the protocol committee during the trial.

6 Participants Patients with inoperable NSCLC stage IIB, III or IV with oligo-metastatic disease and PS 0-2, who are not candidates for standard curative intended radiotherapy. Two general criteria can be used for entry into the protocol: A) The target volume for radiotherapy treatment volume is considered too large for a standard treatment of 66Gy in 33 fractions, considering the expected normal tissue toxicity with a standard treatment plan; or B) The patient is too fragile for standard long-course radiotherapy with 66 Gy.

6.1 Inclusion criteria

* Histologically or cytological confirmed locally advanced, inoperable NSCLC.
* Age ≥18 years.
* Signed informed consent.
* Performance status 0-2.
* Able to comply with study and follow-up procedures.
* Fertile women must have a negative pregnancy test. Fertile men and women must use effective contraception. Fertile women included in the study must use the pill, spiral, depot injection of gestagen, subdermal implantation, hormonal vaginal ring or transdermal patch for the duration of study treatment and one month thereafter.

6.2 Exclusion criteria

* Prior radiotherapy to the thorax, unless there is no significant overlap of current treatment volumes with previous treatment fields.
* Dose plan conforming to protocol planning criteria not possible.
* Uncontrolled metastatic disease.
* Other active malignant disease. 6.3 Enrolment Patients are enrolled prior to initiation of radiotherapy when criteria in 6.1 and 6.2 are met. Patients enrolled are registered in either cohort A or cohort B.

6.4 Evaluations during treatment Patients will be evaluated and treatment toxicity will be registered once during the course of radiotherapy. Adverse Event Registration collected by CTC version 4.0.

6.5 Follow-up Patients will be seen every 3rd month during a follow up period of 24 months and thereafter every 6th month until end of study. During the first 24 months, the patient will be examined every 3rd month with a CT-scan and afterwards twice a year. Lung function test will be performed at 3 months and if needed clinically afterwards. An ECG will be performed at baseline as well as at 3 months.

6.6 Recurrences Local failures are assessed with CT scan of thorax and upper abdomen. All recurrences should be verified by biopsy if possible. Patients with recurrence are kept in the protocol with regards to collection of follow-up data.

7 Complications (Evaluation of toxicity) All complication (side effects) will be evaluated according to the NCI-CTCAE v 4.0 during all follow-up visits.

7.1 Side effects The study is based on an overall de-escalation of dose compared to the standard treatment, so it is generally expected to observe fewer side effects.

7.2 Adverse Event (AE) Any unfavourable and unintended sign or symptom related to the organs in the thorax: the lungs, the pleurae, the oesophagus, the bronchial tree (including the trachea), the heart and the great vessels in the thorax will be reported.

7.3 Serious Adverse Event (SAE) A SAE is an event occurring during any part of the protocol treatment after radiotherapy initiation that results in any of the following: death, a life-threatening experience that requires hospitalization or requires intervention to prevent permanent impairment/damage. All grade 3 or more radiation-induced lung toxicity, esophagitis grade 4, grade 2 pericardial effusion, bronco-pulmonary fistula and oesophagus strictureas recorded using CTC -AE V4 [18]. All SAEs will be evaluated by the local site investigator and reported to the trial management committee.

8 Statistical considerations and planned data analyses This study aims at providing an alternative option to a purely palliative treatment for NSCLC patients with locally advanced disease. Thus the study needs to demonstrate outcomes not considerably inferior to current standard palliative treatment. Current one-year survival for palliative patients in the Danish Oncological Lung Cancer database is 38% (baseline estimate). The investigators assume that the case mix in the current study will consist of somewhat better prognosis patients than the average palliative patient, corresponding to a one-year survival of 48% (i.e. 10%-points better than baseline) in category A patients. In order to establish, with 80% power and one-sided confidence of 95%, that the proposed treatment results in a one-year survival in which is no more than 5%-points inferior to the baseline (i.e. no worse than 33%), 69 patients are needed. In order to account for a loss to follow-up of 10%, the trial plans to accrue 76 patients in category A. Patients included in category B are inherently frail and elderly, with expected worse overall survival than category A patients. Assuming 33% baseline one-year survival and 43% one-year survival for study patients, and maintaining the remainder of the requirements above, 75 category B patients is needed.

The treatment will be considered ineffective if it cannot be concluded that the one year survival rate is no more than 5%-points lower than that of the average palliative patient. Locoregional failure rate will be calculated as a cumulative incidence estimate.

Toxicity, during and after radiotherapy, will be scored using CTC version 4.0 [CTC]. Incidence of acute and late toxicity grade ≥ 3 and grade 5 will be evaluated, with acute toxicity summarized as worst grade during treatment and late toxicity as cumulative incidence of toxicity events.

9 Ethical considerations Patients, who are not candidates for a definitive chemoradiotherapy schedule of 66 Gy in 2 Gy fractions, are most often offered purely palliative intent treatment regimens, either with low dose radiotherapy or chemotherapy. In this study, these patients are offered a radiotherapy schedule with high doses, with an expectation of better survival due to improved local control. This study will be performed according to the appropriate GCP-ICH regulations and in concordance with the Helsinki Declaration (Seoul version, October 2008). Approval from the ethical committee is obtained. The Danish Data Protection Agency is informed. All patients must have agreed to participate by signing the consent form.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytological confirmed locally advanced, inoperable NSCLC.
* Age ≥18 years.
* Signed informed consent.
* Performance status 0-2.
* Able to comply with study and follow-up procedures.
* Fertile women must have a negative pregnancy test. Fertile men and women must use effective contraception. Fertile women included in the study must use the pill, spiral, depot injection of gestagen, subdermal implantation, hormonal vaginal ring or transdermal patch for the duration of study treatment and one month thereafter.

Exclusion Criteria:

* Prior radiotherapy to the thorax, unless there is no significant overlap of current treatment volumes with previous treatment fields.
* Dose plan conforming to protocol planning criteria not possible.
* Uncontrolled metastatic disease.
* Other active malignant disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 12 months
  One year overall survival rate calculated from raditherapy start day

SECONDARY OUTCOMES:
Time to locoregional failure | 60 months
  Cumulative incidence estimate of locoregional failure calculated from radiotherapy start
Incidence of acute toxicity | 6 months
  Incidence of acute toxicity, Dysphagia, cough and pneumonitis evaluated by NCI- CTCAE v 4 grade ≥ 3 and grade 5 will be evaluated, with acute toxicity summarized as worst grade during treatment
Incidence of late toxicity | 60 months
  Incidence of late toxicity grade ≥ 3 and grade 5 will be evaluated using CTC, as cumulative incidence of toxicity events.NCI- CTCAE v 4

CONTACTS AND LOCATIONS:
Overall Officials: Azza A Khalil, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided